CLINICAL TRIAL: NCT06239701
Title: Development of a Lifestyle Physical Activity Intervention to Reduce Risk for Perinatal Cannabis Use - RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34DA055317-02 (NIH)
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either a Fitbit Only Condition, or a Fitbit + A Lifestyle Physical Activity Intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LPA and Fitbit (Experimental): The 12-week LPA+Fitbit intervention consists of 3 components:
  1. In-Person LPA+Fitbit Orientation
  2. Telephone PA counseling sessions.
  3. Fitbit activity tracker.
  Interventions: Behavioral: LPA+Fitbit Intervention
- Only Fitbit (Active Comparator): The Fitbit Only condition will include 3 components:
  1. In-person Fitbit Orientation.
  2. Fitbit Activity Tracker.
  3. Brief Telephone Check-ins.
  Interventions: Behavioral: Fitbit Only

INTERVENTIONS:
Behavioral: LPA+Fitbit Intervention — 1. In-Person LPA+Fitbit Orientation. During an initial, orientation (45 minutes), a study interventionist will provide information regarding the acute and long-term psychological and physical benefits of increasing PA, including prenatally.
  2. Telephone PA counseling sessions. A study interventionist will call participants at weeks 2, 4, 6, 8, and 10 of the intervention for a 20-min telephone session.
  3. Fitbit activity tracker. With participant permission, a Fitbit account (on Fitbit.com) and study-generated password will be created. In doing so, investigators will have access to the participant activity data throughout the intervention. The Fitbit web-based and mobile apps facilitate goal-setting by allowing participants to easily set goals and change these goals at any point. We will customize each participant account to display daily steps and very active minutes, though they will be encouraged to adjust the display according to their preferences.
  Other Names: Women Out Walking
  Arms: LPA and Fitbit
Behavioral: Fitbit Only — 1. In-person Fitbit Orientation. Participants will be given information on the public health guidelines for PA during pregnancy, and as well as how to determine if their PA is moderate-intensity. In addition, interventionists will orient participants to the proper use of the Fitbit tracker and offer tips for self-monitoring step counts with the tracker and on the app.
  2. Fitbit Activity Tracker. Participants will be given the same Fitbit as in the LPA condition. Participants will not be given any specific step count goals to achieve during the 12-week intervention.
  3. Brief Telephone Check-ins. As with the LPA+Fitbit participants, those in the Fitbit Only condition will receive phone calls on weeks 2, 4, 6, 8, 10. These calls will last 5 minutes and be focused entirely on answering any problems related to the Fitbit such as syncing issues, charging the battery, and any other technical problems that may arise. No physical activity counseling will be delivered on these calls.
  Arms: Only Fitbit

SUMMARY:
The overall goal of this pilot study is to develop and preliminarily evaluate an LPA intervention designed to reduce cannabis use during pregnancy.

DETAILED DESCRIPTION:
In the pilot RCT, we will recruit 50 women between 12-22 weeks gestation from an established network of prenatal clinics, and randomly assign eligible women to either a: 1) LPA+Fitbit intervention or 2) Fitbit Only control condition. Similar to our prior trials with pregnant women, the intervention period will be 12 weeks in duration during pregnancy, with follow-ups extending to the end of pregnancy and into the postpartum period. Major assessments will occur at baseline, end of treatment (EOT), and 4 weeks postpartum; we will also conduct brief phone surveys at three points in between the larger assessments. Participants will complete a 7-day period of accelerometry and urine toxicology screens following each major assessments. Birth record abstractions to collect information about specific outcomes (pre-term delivery, low birth weight) will be conducted by trained staff at one month post-birth.

ELIGIBILITY:
Inclusion Criteria:

1. women 18+ years of age
2. 12-25 weeks gestation with a healthy singleton pregnancy
3. medically-cleared by their prenatal provider for moderate intensity physical activity
4. self-report of cannabis use at least once/week in the 3 months prior to the current pregnancy and desire to not engage in prenatal CU
5. current psychological distress as defined by Edinburgh Postnatal Depression Scale score >7 and/or Generalized Anxiety Disorder 7 score >5)
6. English-speaking
7. owns a smartphone to enable use of the Fitbit app
8. current physical activity level does not meet public health recommendations (less than 150 minutes/week moderate intensity physical activity for the past 3 months)
9. expresses interest in reducing or discontinuing CU

Exclusion Criteria:

1. current DSM-5 diagnosis of moderate/severe substance use disorder other than cannabis use disorder or nicotine use disorder
2. use of illicit substances in the last 3 months (other than cannabis)
3. acute psychotic symptoms
4. current or recent suicidality or homicidality
5. current anorexia or bulimia
6. current cognitive impairment
7. physical or medical problems that would not allow safe participation in moderate intensity physical activity
8. has plan to relocate away from the geographic area during the study intervention or assessment period
9. recently started a new form of mental health or substance use treatment within the past 4 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Timeline Follow-back (TLFB) | Baseline to 12-week endpoint
  Interviewer-administered assessment of use of cannabis, alcohol, tobacco, and other drugs
Steps/day | Baseline to 12-week endpoint
  objectively-measured
Activity Minutes/Day | Baseline to 12-week endpoint
  objectively-measured
The Daily Sessions, Frequency & Quantity of Cannabis Use Inventory - Factor 1 | Baseline to 12-week endpoint
  Self-reported cannabis use questionnaire -factor 1: daily sessions
The Daily Sessions, Frequency & Quantity of Cannabis Use Inventory - Factor 2 | Baseline to 12-week endpoint
  Self-reported cannabis use questionnaire - factor 2: frequency
The Daily Sessions, Frequency & Quantity of Cannabis Use Inventory - Factor 3 | Baseline to 12-week endpoint
  Self-reported cannabis use questionnaire - factor 3: age of onset
The Daily Sessions, Frequency & Quantity of Cannabis Use Inventory - Factor 4 | Baseline to 12-week endpoint
  Self-reported cannabis use questionnaire - factor 4: Marijuana quantity
The Daily Sessions, Frequency & Quantity of Cannabis Use Inventory - Factor 5 | Baseline to 12-week endpoint
  Self-reported cannabis use questionnaire - factor 5: Concentrate quantity
The Daily Sessions, Frequency & Quantity of Cannabis Use Inventory - Factor 6 | Baseline to 12-week endpoint
  Self-reported cannabis use questionnaire - factor 6: Edibles quantity
Urine Toxicology Screen | Baseline to 12-week endpoint
  Objective screening for use of cannabis via measurement of THC in urine samples
International Physical Activity Questionnaire | Baseline to 12-week endpoint
  self-report measure of physical activity including minutes/week spent walking, engaging in moderate physical activity, and engaging in vigorous physical activity

SECONDARY OUTCOMES:
Brief COPE | Baseline to 12-week endpoint
  Self-report measure of use of coping strategies; includes 14 2-item scales, each ranging from 2-8. Higher scores indicate increased utilization of a coping strategy.
Marijuana Self-Efficacy Questionnaire | Baseline to 12-week endpoint
  Self-report measure of efficacy for cannabis abstinence; Scores range from 0-100, with higher scores indicating greater use of strategies to reduce marijuana consumption.
Edinburgh Postnatal Depression Screen | Baseline to 12-week endpoint
  Self-report measure of depression severity; scores range from 0-30, with higher scores indicating higher depression
Generalized Anxiety Disorder -7 | Baseline to 12-week endpoint
  Self-report measure of anxiety severity; scores range from 0-21, with higher scoring indicating more anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Battle, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No